CLINICAL TRIAL: NCT00660751
Title: The Role of Central Serotonergic and Adrenergic Systems in the Effectiveness of DNIC (Diffuse Noxious Inhibitory Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, d_yarnitsky, Head of Neurology Department, Rambam Health Care Campus
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: DNIC01CTIL
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Physiology of Serotonergic and Adrenergic systems
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Duloxetine
- 2 (Placebo Comparator)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — SNRIs

SUMMARY:
The role of central serotonergic and adrenergic systems in the effectiveness of DNIC (Diffuse Noxious Inhibitory Control) will be tested before and after taking Duloxetine and Placebo in a double blind study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* age 18-80
* no chronic disease

Exclusion Criteria:

* Subjects who suffer from chronic pain / pain syndrome
* use of anti-depressant or anti-psychotic drugs
* food/ drugs sensitivity
* breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
level of DNIC | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Prof. David Yarnitsky, Principal Investigator
Locations (1):
- Rambam Health Care Campus, Haifa, Israel